CLINICAL TRIAL: NCT07330531
Title: A Drug-drug Interaction Study to Evaluate the Effects of Rifampin Capsules on the Pharmacokinetics of Anaprazole Sodium Enteric-coated Tablets in Healthy Adult Subjects
Brief Title: Drug-drug Interaction Study of Rifampin and Anaprazole Sodium
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanzhu Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3571-DDI-1007
Record Dates: First submitted 2025-12-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Drug-drug Interaction Study
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anaprazole sodium enteric-coated tablets + Rifampin capsules (Experimental): Anaprazole sodium enteric-coated tablets 60 mg once daily (QD) on Day1 and D10, Rifampin capsules 600 mg QD from Day 4-Day11
  Interventions: Drug: Anelazol Sodium Enteric-coated Tablets; Drug: Rifampicin Capsules

INTERVENTIONS:
Drug: Anelazol Sodium Enteric-coated Tablets — 60mg QD
Drug: Rifampicin Capsules — 600mg QD

SUMMARY:
A drug-drug interaction study designed to evaluate the drug-drug interaction between rifampin capsules and anaprazole sodium enteric-coated tablets in healthy adult subjects

DETAILED DESCRIPTION:
This is an open-label, single-center, two-period, single-sequence crossover drug-drug interaction study of rifampin capsules and anaprazole sodium enteric-coated tablets in healthy adult subjects. On Day 1 and Day 10, subjects will orally receive a single 60 mg dose of anaprazole sodium enteric-coated tablets in the morning under fasting conditions. From Day 4 to Day 11, subjects will orally receive 600 mg of rifampin capsules once daily (QD) in the morning under fasting conditions for 8 consecutive days. Specifically, on Day 10, subjects will orally receive both a single 60 mg dose of anaprazole sodium enteric-coated tablets and a 600 mg dose of rifampin capsules in the morning under fasting conditions. Pharmacokinetics will be followed from Day 1 through Day 12.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects aged 18-45 years (including boundary values);
2. Male weight ≥50kg, female weight ≥45kg, body mass index (BMI) in the range of 19-28 kg/m2 (including boundary value);
3. No mental abnormalities, cardiovascular system, nervous system, respiratory system, digestive system, urinary system, history of systemic, endocrine and metabolic abnormalities;
4. The subjects agreed to use effective contraception and had no plans to donate sperm or eggs from the time of trial screening until 6 months after the last dose;
5. The subjects should be able to communicate well with the researchers, understand and comply with the requirements of the study, and understand and sign the informed consent.

Exclusion Criteria:

1. Subjects with a specific allergic history (e.g., urticaria, eczema), an allergic constitution (e.g., allergy to two or more drugs, foods such as milk or pollen), a known allergy to anaprazole sodium or similar drugs, or an allergy to rifampin or its similar antibacterial drugs;
2. During screening, there are clinical significant abnormal results in physical examination, laboratory tests, 12-lead electrocardiogram, chest x-ray examination or abdomen B ultrasound examination;
3. Subjects with a history of drug abuse (including regular use of sedatives, hypnotics, or other addictive substances) within 12 months before screening; or who have used illicit drugs; or test positive in urine drug screening;
4. Subjects who smoked more than 5 cigarettes per day within the 3 months before screening, or who could not stop using any tobacco products during the study;
5. Alcohol breath test positive o regular drinkers within 6 months before screening, drinking more than 14 units per week [1 unit is equivalent to 350 mL of beer (5%), 45 mL of spirits (40%) or 150 mL of wine (12%)];
6. Use any prescription drugs or traditional Chinese medicine within 4 weeks prior to the first dose, or use any OTC drugs or dietary supplements within 2 weeks before the first dose;
7. Participated in other clinical trials and used investigational drugs within 3 months before screening;
8. Those who received live vaccine within 2 weeks before the first dose, or planned to receive live vaccine during the study or within 7 days after the study was completed;
9. Blood donation (including component blood donation) or blood loss of 400 mL within 3 months before screening, or blood transfusion; Blood donation (including component blood donation) or blood loss of 200 mL within 1 month before screening;
10. Have a history of major disease, major surgery, or significant trauma within the 3 months prior to screening, or who plan to undergo surgery during the study;
11. Subjects with dysphagia or a history of gastrointestinal disorders that may affect drug absorption or cause clinically significant symptoms (e.g., gastrectomy or small bowel resection, atrophic gastritis, chronic intestinal diseases, gastrointestinal bleeding, obstruction, etc.), or those with acute gastrointestinal conditions (such as nausea, vomiting, diarrhea, abdominal pain, constipation, etc.) within the week prior to screening;
12. Female subjects during pregnancy and lactation and female subjects of reproductive age who cannot take contraception as required;
13. HBsAg, HCV Ab, Treponema pallidum antibody, HIV Ab test results are positive;
14. Those who have special dietary requirements (including lactose intolerance) and are unable to comply with the provided diet and corresponding regulations;
15. Those who have consumed a special diet (including pitaya, mango, pomelo, and/or xanthine-containing foods, chocolate) and/or have regularly consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, and/or caffeinated beverages (averaging more than 8 cups per day, with each cup being 200 mL) within the 2 weeks prior to the first dose, thereby potentially affecting drug absorption, distribution, metabolism, or excretion;
16. Use of any drug that inhibits or induces hepatic metabolism within 30 days prior to the first dose: Inducer such as barbiturates, carbamazepine, phenytoin sodium, rifamequine; Inhibitors such as cimetidine, cyclosporine, macrolides, verapamil, quinolones, pyrroles, etc.);
17. Those who cannot tolerate blood collection by venipuncture or whose blood vessels are in poor condition;
18. Other subjects deemed unsuitable to participate in the study by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-04 (Estimated); Primary Completion 2026-02-05 (Estimated); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Cmax | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the Cmax of the parent drug and major metabolites of anaprazole sodium in healthy subjects.
AUC0-t | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the AUC0-t of the parent drug and major metabolites of anaprazole sodium in healthy subjects
AUC0-∞ | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the AUC0-∞ of the parent drug and major metabolites of anaprazole sodium in healthy subjects
Tmax | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the Tmax of the parent drug and major metabolites of anaprazole sodium in healthy subjects
t1/2 | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the t1/2 of the parent drug and major metabolites of anaprazole sodium in healthy subjects
CL/F | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the CL/F of the parent drug and major metabolites of anaprazole sodium in healthy subjects
V/F | Day 1 to Day 12
  To assess the effects of multiple oral dose administration of rifampin on the V/F of the parent drug and major metabolites of anaprazole sodium in healthy subjects

SECONDARY OUTCOMES:
The number of subjects with adverse events | From first application of study medication up to 14 days after end of treatment with study medication
  To evaluate the incidence and severity of adverse events (AEs) and serious adverse events (SAEs) of anaprazole sodium administered alone and in combination with rifampin in healthy subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Master, Principal Investigator — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital of Shandong Province, Jinan, Shangdong, China